CLINICAL TRIAL: NCT04206488
Title: A Single-center, Open-label, Fixed-sequence, Study Evaluating the Two-way Drug-drug Interaction Between JNJ-70033093 and Digoxin in Healthy Subjects
Brief Title: A Study of JNJ-70033093 and Digoxin in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108712; 70033093THR1001 (Other: Janssen Research & Development, LLC); 2019-003783-46 (EudraCT Number)
Record Dates: First submitted 2019-12-18; First posted 2019-12-20 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Healthy
MeSH Terms: interventions — milvexian; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-70033093 + Digoxin (Experimental): Participants will receive JNJ-70033093 as oral capsules (Treatment A) in Period 1, followed by digoxin tablets as loading dose and maintenance doses (Treatment B) in Period 2, and then digoxin tablets along with JNJ-70033093 (Treatment C) in Period 3. There will be a washout period of minimum 5 days (and maximum 7 days) between the last dosing day of Period 1 and the first dosing day of Period 2. There is no washout between Periods 2 and 3 (that is, the last day of Treatment B is to be followed by the first day of Treatment C).
  Interventions: Drug: JNJ-70033093; Drug: Digoxin

INTERVENTIONS:
Drug: JNJ-70033093 — Participants will receive JNJ-70033093 orally.
  Other Names: BMS-986177
Drug: Digoxin — Participants will receive digoxin orally.
  Other Names: Lanoxin

SUMMARY:
The purpose of this study is to evaluate the potential pharmacokinetic (PK) interaction between JNJ-70033093 and digoxin in healthy participants after single dose administration and at steady state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, medical history, vital signs, Electrocardiogram (ECG), and laboratory test results, including serum chemistry, blood coagulation, hematology, and urinalysis performed at screening. If there are abnormalities, the investigator may decide that the abnormalities or deviations from normal are not clinically significant, in which case the participant may be included. This determination must be recorded in the participant's source documents and initialed by the investigator
* Normal renal function at screening as evidenced by an estimated glomerular filtration rate (eGFR) of greater than or equal to (>=) 90 milliliter per minute (mL/min) per 1.73 meter square (m^2) calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula
* A woman of childbearing potential must have a negative serum beta human chorionic gonadotropin (beta-hCG) test at screening and a negative urine (beta-hCG) test on Day -1 of Period 1
* Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies. Before screening, a woman must either be: a) Not of childbearing potential b) Of childbearing potential c) Women must have no history of excessive menstrual bleeding or hemorrhage following pregnancy delivery
* Body mass index (BMI; weight [kilogram {kg}] per height square (height^2 [meter^2]) between 18.0 and 30.0 kilogram per meter square (kg/m^2) (inclusive), and body weight not less than 55 kg
* A 12-lead ECG consistent with normal cardiac conduction and function at screening and on Day 1 of Period 1, including: a) Sinus rhythm, b) Heart rate between 55 and 90 beats per minute (bpm), c) Corrected QT (QTc) interval of less than or equal to (<=) 450 milliseconds (ms) for male participants and <= 470 ms for female participants (QT interval will be corrected for heart rate using the Fridericia correction, d) QRS interval of less than (<) 110 ms, e) PR interval <200 ms, f) Morphology consistent with healthy cardiac conduction and function

Exclusion Criteria:

* Participant is a woman who is pregnant, breastfeeding, or planning to become pregnant during this study or within 34 days after the last study drug administration
* History of or current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, gastrointestinal disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* History of clinically significant ECG abnormalities, sinus node disease, or incomplete atrioventricular (AV) block or a family history of prolonged QT interval syndrome
* Positive blood screen for hepatitis C virus antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) type 1 and type 2 antibody
* Use of any prescription or nonprescription medication (including vitamins and herbal supplements), except for oral contraceptives, hormonal replacement therapy (HRT), and paracetamol, within 14 days before the first dose of the study drug is scheduled
* Received an experimental drug/placebo or used an experimental medical device within 3 months or within a period less than 5 times the drug's half-life (whichever is longer) prior to the planned first dose of study drugs or is enrolled in an investigational study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Geometric Mean Ratio of Treatment C (JNJ-70033093 + Digoxin) Relative to Treatment A (JNJ-70033093) | Up to Day 21
  Cmax is the maximum observed plasma concentration. Cmax geometric mean ratio of Treatment C (JNJ-70033093 + digoxin) relative to Treatment A (JNJ-70033093) will be reported to assess the effect of digoxin on the pharmacokinetics (PK) of JNJ-70033093.
Cmax Geometric Mean Ratio of Treatment C (JNJ-70033093 + Digoxin) Relative to Treatment B (Digoxin) | Up to Day 21
  Cmax is the maximum observed plasma concentration. Cmax geometric mean ratio of Treatment C (JNJ-70033093 + Digoxin) relative to Treatment B (digoxin) will be reported to assess the effect of JNJ-70033093 on the PK of digoxin.
Area Under the Plasma Concentration-time Curve from Time 0 to 24 Hours Postdose (AUC [0-24 hours]) Geometric Mean Ratio of Treatment C (JNJ-70033093 + Digoxin) Relative to Treatment A (JNJ-70033093) | Up to 24 hours postdose
  AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours postdose. AUC (0-24) geometric mean ratio of Treatment C (JNJ-70033093 + digoxin) relative to Treatment A (JNJ-70033093) will be reported to assess the effect of digoxin on the PK of JNJ-70033093.
AUC (0-24) Geometric Mean Ratio of Treatment C (JNJ-70033093 + Digoxin) Relative to Treatment B (Digoxin) | Up to 24 hours postdose
  AUC (0-24) is the area under the plasma concentration-time curve from time zero to 24 hours postdose. AUC (0-24) geometric mean ratio of Treatment C (JNJ-70033093 + digoxin) relative to Treatment B (digoxin) will be reported to assess the effect of JNJ-70033093 on the PK of digoxin.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a Measure of Safety and Tolerability | Up to 63 Days
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product does not necessarily have a causal relationship with the treatment. Therefore, it can be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not related to that medicinal product.
Number of Participants with Vital Sign Abnormalities as a Measure of Safety and Tolerability | Up to 63 Days
  Number of participants with vital sign (tympanic temperature, resting [supine] pulse rate, and blood pressure) abnormalities will be reported.
Number of Participants with 12-lead Electrocardiogram (ECG) Abnormalities as a Measure of Safety and Tolerability | Up to 63 Days
  Number of participants with 12-lead ECG abnormalities will be reported.
Number of Participants with Laboratory Abnormalities as a Measure of Safety and Tolerability | Up to 63 Days
  Number of participants with laboratory abnormalities (hematology, coagulation tests, clinical chemistry, and urinalysis) will be reported.
Percent Change From Baseline in Activated Partial Thromboplastin Time (aPTT) | Baseline up to Day 21
  Percent change from baseline in aPTT will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency